CLINICAL TRIAL: NCT01742845
Title: Ultrasound-guided Intermediate Cervical Block Versus Superficial Cervical Block for Carotid : a Randomised Controlled Trial
Brief Title: Ultrasound-guided Intermediate Cervical Block Versus Superficial Cervical Block for Carotid Endarterectomy (CERVECHO)
Acronym: CERVECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P/2010/107
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Carotid Atherosclerosis; Regional Anaesthesia Morbidity
Keywords: Ultrasound-guided; regional anaesthesia; Cervical block
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Active Comparator): landmark-based superficial cervical block is used. After insertion of the needle superficially below the skin, 20 to 30 ml of 4.75 mg/ml ropivacaine are injected fan-like in the subcutaneus plane.
  Interventions: Other: landmark based superfical ropivacaine 4.75 mg/ml injection
- echo group (Experimental): ultrasound-guided intermediate cervical block was performed. The probe is placed perpendicular to the skin, in the horizontal plane at the C3-C4 level. Needle is inserted in-plane. 10 ml ropivacaine 4.75mg/ml are injected under ultrasound control, 5 ml injected when needle is withdrawn under ultrasound control, 5 ml in the subcutaneous plane.
  Interventions: Other: Ultrasound-guided administration of ropivacaine 4.75 mg/ml

INTERVENTIONS:
Other: Ultrasound-guided administration of ropivacaine 4.75 mg/ml
  Arms: echo group
Other: landmark based superfical ropivacaine 4.75 mg/ml injection
  Arms: control group

SUMMARY:
The aim of this prospective, randomised, controlled study is to compare the efficacy of ultrasound-guided intermediate cervical block to superficial block for carotid endarterectomy.

Patients scheduled for carotide endarterectomy under regional anaesthesia (ropivacaine 4.75 mg/ml) are randomised into 2 groups according to the technique of anaesthesia performed: superficial cervical block (Control group) or, ultrasound guided intermediate cervical block (Echo group). Main outcome is cervical block success, defined by surgery performed under regional anaesthesia without supplemental topical lidocaine. Secondary outcomes are rate of conversion to general anaesthesia, total dose of supplemental topical lidocaine and block-related complications.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for elective carotid artery endarterectomy under regional anaesthesia

Exclusion Criteria:

* indication for general anaesthesia
* known bleedind diathesis
* past medical allergy to local anaesthesic
* severe chronic pulmonary disease
* contralateral diaphragmatic motion abnormalities
* previous cervical ipsilateral surgery
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
cervical block success | surgery time
  carotid artery endarterectomy performed under regional anaesthesia without supplemental topical lidocaine.

SECONDARY OUTCOMES:
percentage of conversion to general anaesthesia | surgery time
  conversion to general anaesthesia for insufficient analgesia

OTHER OUTCOMES:
percentage of patient needing intraoperative systemic analgesia or sedation | anaesthesia time
  if patient related pain in spite of supplemental local anaesthesic. sedation/analgesia let to the discretion of the anesthesist in the operating room
amount of local anaesthesic used to performed the block | surgery time
regional anaesthesia-related complications | 7 postoperative days
  Horner syndrom, facial paralysis, cough, phrenic paralysis
surgery related complications | 7 postoperative days
  hematoma, stroke, bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Petit, MD, Principal Investigator — CHRU Besançon; Sebastien Pili-Floury, MD PhD, Principal Investigator — CHRU Besançon
Locations (1):
- Centre Hospitalier universitaire de Besançon, Besançon, France